CLINICAL TRIAL: NCT02074878
Title: A Phase IB Study of Crizotinib (XALKORI) and Sunitinib (SUTENT) in Metastatic Breast Cancer
Brief Title: CRIZENT: Crizotinib and Sunitinib in Metastatic Breast Cancer
Acronym: CRIZENT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual so the study was halted on May 16, 2017.
Sponsor: Mothaffar Rimawi (Other)
Responsible Party: Sponsor-Investigator, Mothaffar Rimawi, Medical Director, Baylor Breast Care Center
Organization: Baylor Breast Care Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33624
Record Dates: First submitted 2013-12-17; First posted 2014-02-28 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic; Crizotinib; Sunitinib; Xalcori; Sutent
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Crizotinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crixotinib 200 mg and Sunitinib Cohort 1 (Experimental): Crizotinib 200mg, twice daily and Sunitinib 25.0mg once daily
  Interventions: Drug: Crixotinib 200 mg and Sunitinib Cohort 1
- Crixotinib 250 mg and Sunitinib Cohort 2 (Experimental): Crizotinib 250 mg, twice daily with Sunitinib 25.0 mg once a day
  Interventions: Drug: Crixotinib 250 mg and Sunitinib Cohort 2
- Crizotinib & Sunitinib 37.5 mg Cohort 3 (Experimental): Crizotinib 250 mg, twice daily with Sunitinib 37.5 mg once a day
  Interventions: Drug: Crizotinib & Sunitinib 37.5 mg Cohort 3

INTERVENTIONS:
Drug: Crixotinib 200 mg and Sunitinib Cohort 1 — Crizotinib 200 mg, twice daily with Sunitinib 25.0 mg once a day
  Other Names: Crizotinib (Xalkori) 200 mg twice daily; Sunitinib (Sutent) 25.0 mg once a day
  Arms: Crixotinib 200 mg and Sunitinib Cohort 1
Drug: Crixotinib 250 mg and Sunitinib Cohort 2 — Crizotinib 250 mg, twice daily with Sunitinib 25.0 mg once a day
  Other Names: Crixotinib (Xalkori) 250; Sunitinib (Sutent) 25.0
  Arms: Crixotinib 250 mg and Sunitinib Cohort 2
Drug: Crizotinib & Sunitinib 37.5 mg Cohort 3 — Crizotinib 250 mg, twice daily with Sunitinib 37.5 mg once a day
  Other Names: Crizotinib (Xalkori) 250 mg; Sunitinib (Sutent) 37.5 mg
  Arms: Crizotinib & Sunitinib 37.5 mg Cohort 3

SUMMARY:
This is a Phase 1 Trial. Crizotinib is a medication that is taken by mouth. It has shown that it can help slow down or stop the growth of tumor cells. The marketing name of the drug is "Xalkori". It has been approved by the FDA (Food and Drug Administration) to treat other types of metastatic cancer, but the investigators believe it may be helpful to treat breast cancer as well.

Sunitinib is the other medication used in the study. It is also taken by mouth in the form of a capsule. The marketing name of this drug is "Sutent". It too has been approved by the FDA to treat other types of cancer, but not for breast cancer.

In this study the investigators will be combining both of these two treatments, but at different doses.

One third of the patients will take Crizotinib 200 mg, twice daily with Sunitinib 25.0 mg once a day.

One third of the patients will take Crizotinib 250 mg, twice daily with Sunitinib 25.0 mg once a day, and One third of the patients will take Crizotinib 250 mg, twice daily with Sunitinib 37.5 mg once a day.

DETAILED DESCRIPTION:
This study will determine the safety and tolerability of the combination of crizotinib and sunitinib in the treatment of Metastatic Breast Cancer and help to establish the maximum tolerated dose for future phase II studies of the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up.
2. Age of at least 18 years
3. Histologically confirmed diagnosis of stage IV, HER2 negative breast cancer.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Patients must have failed two lines of systemic therapy for breast cancer. Patients who are hormone receptor positive must have failed at least one line of hormonal therapy AND one line of chemotherapy in the metastatic setting.
6. Life expectancy of 6 months or more.
7. Liver function (ALT, AST, alkaline phosphatase, total bilirubin) and kidney function tests (BUN, creatinine) less than 2.5 times the upper limit of normal. In patients with liver metastasis, liver function tests should be less than 5 times the upper limit of normal.
8. Adequate blood counts (Hemoglobin greater than/equal to 10, WBC greater than/equal to 3.0, platelets greater than/equal to 100).
9. The patient has normal thyroid function tests (TSH, free T4) as defined by the testing laboratory, a test abnormality that is asymptomatic and does not warrant medical intervention, or a pre-existing thyroid disorder that is controlled on medical treatment.
10. Negative pregnancy test (BHCG) within 14 days of study drug initiation for pre- or perimenopausal subjects with an intact uterus.

Exclusion Criteria:

1. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
2. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational products.
3. Presence of uncontrolled infection.
4. Corrected QT interval (QTc) > 480 msecs using Bazett's formula
5. History of any one or more of the following cardiovascular conditions within the past 6 months: - Cardiac angioplasty or stenting - Myocardial infarction - Unstable angina - Coronary artery bypass graft surgery - Symptomatic peripheral vascular disease - Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
6. Poorly controlled hypertension (defined as systolic blood pressure [SBP] of > 150 mmHg or diastolic blood pressure [DBP] of > 90 mmHg).
7. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism, or untreated deep venous thrombosis (DVT) within the past 6 months. Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
8. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
9. Evidence of active bleeding or bleeding diathesis.
10. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
11. Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks prior to first dose of study drug.
12. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
13. Patients previously treated with sunitinib or crizotinib.
14. History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma of the skin.
15. Concurrent use of: - Potent CYP3A4 inhibitors: ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, amprenavir, indinavir, nelfinavir, delavirdine and voriconazole. - CYP3A4 inducers: rifampin, rifabutin, rifapentin, phenobarbital, phenytoin, carbamazepine, St. John's Wort, and dexamethasone. Use of dexamethasone for study premedication is allowed. - Grapefruit and grapefruit juice. (Note: Alternative therapies should be used when available. If use of a potent CYP3A4 inhibitor or inducer is necessary, this must be approved by the principal investigator and documented in source documents).
16. History of receiving any investigational treatment within 28 days of study medication initiation.
17. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, thyroid, or metabolic disease; wound healing disorders; ulcers; or bone fractures).
18. Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of the treatment drugs in the patients that are taking it. | 1 year
  To determine the tolerability of the combination of crizotinib and sunitinib in the treatment of women with metastatic breast cancer (MBC). - This is done by identifying the maximum tolerated dose (MTD) for future phase II studies of the combination of crizotinib and sunitinib.

SECONDARY OUTCOMES:
Changes that occur in tumor tissue before treatment and after treatment. | 2 years
  Assess the clinical activity of the combination regimen in patients with MBC. - This is done by performing exploratory correlative studies on tissue acquired from accessible metastatic lesions based on serial biopsies performed at baseline and recording changes in biomarker levels between responders vs. non-responders.
Laboratory results to make sure the treatment is safe. | 1 year
  Safety and toxicity parameters will be summarized using descriptive statistics. All patients who received any amount of study drugs will be included in the safety analysis. Safety analyses will include summaries of adverse event rates (both frequency and incidence tables), baseline laboratory parameters and changes from baseline, frequency of CTCAE toxicity grades for both laboratory and non-laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Lester and Sue Smith Breast Center, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No